CLINICAL TRIAL: NCT03628963
Title: Personalize Concerto: A Study Protocol for Optimizing Patient Usability Experience With an eHealth Platform for Embedded, Coordinated and Efficient Healthcare
Brief Title: Optimizing Patient Usability Experience for Chronic Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Collaborators: Concerto Health Group Montréal, Qc, Canada (Unknown); International Business Machines (IBM) (Industry); Vrije Universiteit Brussel, Jette, Belgium (Unknown); Université de Montréal (Other); Haute Ecole de Santé Vaud (HESAV), Lausanne, Switzerland (Unknown)
Responsible Party: Principal Investigator, Marie-Pierre Gagnon, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-067/01-06-2018
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Chronic Disease
Keywords: Diabetes; hypertension; dyslipidemia
MeSH Terms: conditions — Chronic Disease; Diabetes Mellitus; Hypertension; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Two Family Medicine Groups (FMG) from the same health region but covering distinct areas have been selected as the clusters. The FMGs will be randomily selected for the experimental (CONCERTO+) or control (usual care) group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concerto+ (Intervention group) (Experimental): Patients with two or more targeted chronic diseases (diabetes, hypertension, dyslipidemia) and who had three or more visits in the last 12 months will use Concerto+ application during 6 months.
  Interventions: Device: Concerto+
- Usual care (Control group) (No Intervention): Patients with two or more targeted chronic diseases (diabetes, hypertension, dyslipidemia) and who had three or more visits in the last 12 months will not use the application Concerto+ but receive usual care from FMG.

INTERVENTIONS:
Device: Concerto+ — a user-centered, multifunctional and personalized eHealth platform
  Arms: Concerto+ (Intervention group)

SUMMARY:
The study aims to develop a module of an eHealth platform, do a feasibility study through a pilot cluster randomized control trial and assess the scalability of the solution.

DETAILED DESCRIPTION:
Multimorbidity increases care needs and primary care use among people with chronic diseases (1). The Concerto Health Program (CHP) has been developed to optimize chronic disease management in primary care services. However, in its current version, the CHP primarily targets clinicians and does not aim to respond directly to the needs of patients and their informal caregivers for chronic disease management . This project aims to develop, implement and evaluate a user-centered, multifunctional and personalized eHealth platform (CONCERTO+) to promote a more active patient role in chronic disease management and decision-making through three phases.

For phase1: A first prototype will be developed by the design and technology teams, in close collaboration with researchers, health professionals and patient representatives who will identify the functionalities to include in the CONCERTO+ solution.

The Phase 2 of the project will consist in a feasibility study based on a pilot cluster randomized clinical trial (c-RCT) where patients with chronic diseases from a primary healthcare practice will receive CONCERTO+ and be compared to patients from a control practice receiving usual care.

For Phase 3, the analysis of CONCERTO+ potential for scaling-up will be done by documenting factors and conditions associated with the sustainability and scaling-up of the solution. To do so, the investigators will conduct: 1) two focus groups with patients and informal caregivers who participated in the study (one with the experimental group and one with the control group, each group gathering between eight and twelve participants); 2) semi-structured individual interviews with health professionals at the two study sites, as well as with health care managers, information officers, and representatives of the Ministry of Health and Social Services.

ELIGIBILITY:
Inclusion Criteria:

* Having one or more targeted chronic diseases (diabetes, hypertension, dyslipidemia)
* had 3 or more visits in the last 12 months
* having an interest in health and technologies,
* be able to read and speak in French

Exclusion Criteria:

* Majors whose incapacity has been recognised judically

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Patient Activation | 6 months
  The Patient Activation Measure -13 (2) is built on patient knowledge, skills and confidence that are directly targeted by the intervention and is associated to their activation level. Patients who are more activated have better health outcomes. Patients answer to a survey of 13 questions with the following scoring for each answer:
  Strongly disagree = 1; Disagree = 2; Agree = 3; strongly agree = 4
  The score of the activation level obtained (between 0 and 100) shows the degree of ability to manage their health with confidence according to the following scale ranges:
  1. Not believing that activation is important (≤ 47)
  2. Lack of knowledge or confidence to take action (47.1 - 55.1)
  3. Beginning to take action (55.2 - 67)
  4. Taking action (≥ 67.1).

SECONDARY OUTCOMES:
Process of care | 9 months
  The effects of the use of Concerto + will be assessed and measured, using an adapted version of a survey from Glasgow et al. [3] and validated in the previous CHP (Concerto Health Program) assessment. Patients answer to a questionnaire six months after the use of Concerto+. 5 scales based on the key components of Concerto + are defined, and each scale include items: Solving-problems/Advices (4 items), Delivery System Design/Decision support (3 items), Goal Setting/Tailoring (5 items), Follow-up/coordination (5 items), Overall care (9 items). Items are scored on a 5-point scale ranging from 1 (Almost never) to 5 (Almost always), through following subscales 2 (Generally not); 3 (Sometimes); 4 (Most of the time). Higher scores from the assessment survey have better effects in care outcomes.
Acceptability | 9 months
  The acceptability of the device Concerto+ will be assessed by patient and informal caregiver, at the end of the intervention with:
  1. A short survey adapted from the Technology Acceptance Model [4] that includes 3 criteria (perceived ease of use, perceived usefulness, behavioral intention to use) with the following scoring: Strongly disagree = 1; Disagree = 2; Agree = 3; strongly agree = 4. Higher scores rates have a better acceptance of the use of Concerto+.
  2. The use of CONCERTO+ that will be measured by logs (Tests numbers, emergency visits, hospitalizations).

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Pierre Gagnon, Ph.D, Principal Investigator — Faculty of Nursing, Université Laval, Quebec City, QC, Canada
Locations (1):
- Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fortin M, Contant E, Savard C, Hudon C, Poitras ME, Almirall J. Canadian guidelines for clinical practice: an analysis of their quality and relevance to the care of adults with comorbidity. BMC Fam Pract. 2011 Jul 13;12:74. doi: 10.1186/1471-2296-12-74. PMID 21752267
- [Background] Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005 Dec;40(6 Pt 1):1918-30. doi: 10.1111/j.1475-6773.2005.00438.x. PMID 16336556
- [Background] Glasgow RE, Wagner EH, Schaefer J, Mahoney LD, Reid RJ, Greene SM. Development and validation of the Patient Assessment of Chronic Illness Care (PACIC). Med Care. 2005 May;43(5):436-44. doi: 10.1097/01.mlr.0000160375.47920.8c. PMID 15838407
- [Background] Davis, F.D., Perceived usefulness, perceived ease of use, and user acceptance of information technology. MIS quarterly, 1989: p. 319-340
- [Derived] Gagnon MP, Ndiaye MA, Larouche A, Chabot G, Chabot C, Buyl R, Fortin JP, Giguere A, Leblanc A, Legare F, Motulsky A, Sicotte C, Witteman HO, Kavanagh E, Lepinay F, Roberge J, Deletroz C, Abbasgholizadeh-Rahimi S. Optimising patient active role with a user-centred eHealth platform (CONCERTO+) in chronic diseases management: a study protocol for a pilot cluster randomised controlled trial. BMJ Open. 2019 Apr 2;9(4):e028554. doi: 10.1136/bmjopen-2018-028554. PMID 30944143